CLINICAL TRIAL: NCT06523270
Title: Advanced Imaging Holistic Omics Biobank
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Other Study IDs: AIMOMICS-BANK
Record Dates: First submitted 2024-07-18; First posted 2024-07-26 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Oncologic Disorders; Neurologic Disorder; Pulmonary Disease; Cardiovascular Diseases
MeSH Terms: conditions — Nervous System Diseases; Lung Diseases; Cardiovascular Diseases | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- prospective cohort: All adult (≥18 y.o) subjects (until 50000 individuals) presenting to the U.O of Radiologia DiMer "Advanced Imaging for Personalized Medicine" to be submitted to imaging study on advanced scanner
  Interventions: Radiation: Computed Tomography (CT) using Photon Counting CT scanner (Neaotom Alpha, Siemens) and Magnetic Resonance (MRI)

INTERVENTIONS:
Radiation: Computed Tomography (CT) using Photon Counting CT scanner (Neaotom Alpha, Siemens) and Magnetic Resonance (MRI) — All adult (≥18 y.o) subjects (until 50000 individuals) presenting to the U.O of Radiologia DiMer "Advanced Imaging for Personalized Medicine" to be submitted to imaging study on advanced scanner

SUMMARY:
Imaging methods today represent the pillar of prevention, diagnosis, patients monitoring and treatment. Improvement in technology led the development of increasingly high-performance scanners whose potential has not yet been fully explored. In particular, recently introduced photon counting CT scanner and new high filed MRI offers a lake of latent information derived from the images (e.g. spectral data from CT) of potentially great interest and potentially able to provide new insight but that are currently mostly unexplored .These features are also called "opportunist features" because they are in each exam and can be freely derived from images without changing the study protocol used for clinical practice examination but extracted a posteriori from the images representing a precious source of deep characterization of the patients, equally or even more than a genomic analysis, with possible high relevance in the field of screening and prevention, being able to contribute to defining signatures indicating a particular risk of remotely developing a specific pathological condition. The prospective collection of clinical and imaging data from subjects undergoing diagnostic tests with advanced technology has the potential to increase knowledge of the pathophysiological mechanisms of different pathological conditions, to explore and validate the diagnostic-predictive value of opportunistic features not currently used in practice clinical, to increase the diagnostic and prognostic accuracy of CT and MRI examinations and to provide a unique pool for scientific research. Previous relevant experience was conducted in the United Kingdom (UK biobank) where data from over 500,000 patients have been collected in the last 10 years, providing an enormous pool for spontaneous and funded scientific research. This project (UK biobank), although of enormous scientific value, is currently obsolete in terms of the imaging technology used.

DETAILED DESCRIPTION:
The present study is a observational prospective single center study aimed to build a large-scale multiomic database of patients submitted to advanced imaging study performed Photon Counting TC (Neaotom Alpha, Siemens) and 3T Magnetic Resonance Imaging (MR 7700, Philips).

Consecutive adult patients submitted to the aforementioned imaging modality will be enrolled.

For the enrolled patients imaging raw data will be stored additionally to conventional images, routinely stored for legal requirements.

At the time of enrollment clinical, demographic and lab test will be collected as well as results from genetic test if available, and related previous imaging study (e.g. mammography in patients submitted to whole body MRI or breast MRI, colonscopy in patients submitted to abdominal CT or MRI).

For patients candidate to imaging examination using contrast media at the time of needle position for contrast administration a blood sample will be collected for lab test analysis.

In case of imaging, clinical and laboratory examination performed at OSR, these data will be automatically collected.

Annual update is required by the study with the questionnaires and interviews performed with in site clinical visit, telehealth or whenever no one of the previous method is feasible with telephonic call.

During the annual follow-up, clinical, lab test and imaging data will be collected.

If patients perform annual check-up at OSR, it will ask to automatically update patients' record with those information and results.

Data collected and updated will be chosen according to the patients specific risk profile and the clinical indication to perform III level imaging.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (>18 y.o.) submitted to Computed Tomography (CT) using Photon Counting CT scanner (Neaotom Alpha, Siemens) and Magnetic Resonance (MRI) exams acquired with 3T scanner (MR 7700, Philips) for examination required for clinical practice or for clinical trials at the IRCCS San Raffaele Hospital who signe an Informed Consent authorizing data collection.

Exclusion Criteria:

* Absent informed consent signed

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult (≥18 y.o) subjects (until 50000 individuals) presenting to the U.O of Radiologia DiMer "Advanced Imaging for Personalized Medicine" to be submitted to imaging study on advanced scanner
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2024-09-15 (Actual); Primary Completion 2034-09-15 (Estimated); Study Completion 2034-09-15 (Estimated)

PRIMARY OUTCOMES:
a large scale multiomics archive of patients submitted to advanced imaging studies to support a wide range of research intended to identify imaging signature able to improve the prevention, diagnosis and treatment of disease | Follow-up collection yearly for 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Background] Petralia G, Koh DM, Attariwala R, Busch JJ, Eeles R, Karow D, Lo GG, Messiou C, Sala E, Vargas HA, Zugni F, Padhani AR. Oncologically Relevant Findings Reporting and Data System (ONCO-RADS): Guidelines for the Acquisition, Interpretation, and Reporting of Whole-Body MRI for Cancer Screening. Radiology. 2021 Jun;299(3):494-507. doi: 10.1148/radiol.2021201740. Epub 2021 Apr 27. PMID 33904776
- [Background] Summers P, Saia G, Colombo A, Pricolo P, Zugni F, Alessi S, Marvaso G, Jereczek-Fossa BA, Bellomi M, Petralia G. Whole-body magnetic resonance imaging: technique, guidelines and key applications. Ecancermedicalscience. 2021 Jan 7;15:1164. doi: 10.3332/ecancer.2021.1164. eCollection 2021. PMID 33680078
- [Background] Hagen F, Soschynski M, Weis M, Hagar MT, Krumm P, Ayx I, Taron J, Krauss T, Hein M, Ruile P, von Zur Muehlen C, Schlett CL, Neubauer J, Tsiflikas I, Russe MF, Arnold P, Faby S, Froelich MF, Weiss J, Stein T, Overhoff D, Bongers M, Nikolaou K, Schonberg SO, Bamberg F, Horger M. Photon-counting computed tomography - clinical application in oncological, cardiovascular, and pediatric radiology. Rofo. 2024 Jan;196(1):25-35. doi: 10.1055/a-2119-5802. Epub 2023 Oct 4. English, German. PMID 37793417